CLINICAL TRIAL: NCT00539786
Title: Clinical Usefulness of Proton Pump Inhibitor Test for Identifying Gastroesophageal Reflux Disease in Patients With Extraesophageal Symptoms
Brief Title: The Proton Pump Inhibitor (PPI) Test for the Extraesophageal Manifestation of GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Poong-Lyul Rhee, Professor, Samsung Medical Center
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-03-071
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Patients with extraesophageal manifestation of gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Proton Pump Inhibitors; Rabeprazole

INTERVENTIONS:
Drug: Proton pump inhibitor (rabeprazole) — Patients receives rabeprazole 20mg AM and 20mg PM for 14 days

SUMMARY:
PPI test;empirical trial with high-dose proton-pump inhibitors (PPIs) has been shown to be a sensitive tool for diagnosing patients with GERD. However, this diagnostic strategy has not been well established in patients with extraesophageal manifestation of GERD. In this study, we aim to see the relevance of PPI test in diagnosing GERD in patients with extraesophageal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extraesophageal manifestation symptoms of GERD

Exclusion Criteria:

* laryngeal, pharyngeal, liver, lung, renal, or hematological disorders
* a history of gastrointestinal surgery, and a history of connective tissue disorders.
* patients with duodenal or gastric ulcers as well as other significant lesions, such as gastric cancer, esophageal cancer, or subepithelial tumors more than 1 cm observed on the upper endoscopy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Symptom responders after PPI trials | 2 weeks after PPI trials

CONTACTS AND LOCATIONS:
Overall Officials: Poong-Lyul Rhee, MD. Ph.D, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Gangnam-gu, South Korea